CLINICAL TRIAL: NCT01997151
Title: Promoting Health During Pregnancy: A Multiple Behavior Computer Tailored Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Principal Investigator, Leanne Mauriello, Vice President of Research and Product Development, Pro-Change Behavior Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRANT10236132; 5R44DP001115-03 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Life Stress; Smoking Cessation; Poor Nutrition
MeSH Terms: conditions — Stress, Psychological; Smoking Cessation; Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Pregnancy: Step by Step (Experimental): Pregnant women interacted with a multiple behavior change iPad- delivered program at federally funded health centers. The 20-30 minute program offered onscreen assessments of Transtheoretical Model strategies of change, and then provided individually tailored feedback messages matched to their readiness to change for relevant target behaviors. The program addressed smoking cessation and relapse prevention, stress management, and fruit and vegetable consumption. The feedback screens were interactive and engaging. The messages were written at a 4th-5th grade level and were reviewed for multicultural relevancy. Participants in the treatment group interacted with the program up to 3 times during pregnancy. A printed multiple behavior change guide also was distributed. All program components are available in English and Spanish.
  Interventions: Behavioral: Healthy Pregnancy: Step by Step
- Usual Care (No Intervention): Pregnant women received regular prenatal care as delivered by the health care center from where they were receiving care. Standard informational March of Dimes brochures related to the target behaviors were distributed to usual care participants.

INTERVENTIONS:
Behavioral: Healthy Pregnancy: Step by Step
  Arms: Healthy Pregnancy: Step by Step

SUMMARY:
This program of research tested the effectiveness of an iPad delivered multiple behavior intervention grounded in the Transtheoretical Model of Behavior Change for pregnant women. It was hypothesized that the intervention would reduce the number of health behavior risks reported by pregnant women in the treatment group. The target behaviors of the intervention are smoking cessation and relapse prevention, stress management, and fruit and vegetable consumption.

DETAILED DESCRIPTION:
Promoting health behaviors during pregnancy has tremendous public health significance. Poor health behaviors are associated with pregnancy complications, birth outcomes, and the health of the child. They influence infant birthweight, premature birth, and infant mortality rates, all of which continue to be public health concerns, reflected in the goals of Healthy People 2020.

Pregnant women, particularly those from under-served populations, often have a multitude of health behavior risks that threaten positive pregnancy and birth outcomes, as well as the future health of mother and baby. Pregnancy offers a window of opportunity for behavioral intervention. The immediate health risk for the baby motivates most pregnant women to at least consider changing their behavior. Furthermore, the regular and continual medical care that most pregnant women receive allows optimal access for intervention. The circumstance of pregnancy can be used as a teachable moment to better the future health of women and children.

The primary goals of this study were to complete and enhance the development of an iPad delivered intervention and to assess the efficacy in a randomized clinical trial involving pregnant women from three federally-funded community health centers that treat under-served populations. Using interactive technology, users complete onscreen assessments and receive individually tailored feedback messages on key behavior change strategies identified by the Transtheoretical Model of Behavior Change and matched to their stage of readiness for each behavior. Supplemental intervention components were created including printed feedback reports, a multiple behavior stage-based manual, and Spanish versions of all intervention materials. This intervention offers a cost-effective, science based, and easily deliverable solution to improve multiple health behaviors, and overall health and well-being, of populations of pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Speak and read either English or Spanish
* Consent to the research.

Exclusion Criteria:

* More than 18 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in number of health behavior risks from Baseline at third trimester, 1 month post delivery, and 4 months post delivery | Third trimester of pregnancy, 1 month post delivery, 4 months post delivery
  Health risks were defined as not meeting criteria for smoking (not smoking), fruit and vegetable consumption (eating at least 5 servings a day), and stress management (effectively managing stress).
Change in number of minutes spent on stress management each day from Baseline at third trimester, 1 month post delivery, and 4 months post delivery | Third trimester of pregnancy, 1 month post delivery, 4 months post delivery
Change in number of servings of fruits and vegetables consumed each day from Baseline at third trimester, 1 month post delivery, and 4 months post delivery | Third trimester of pregnancy, 1 month post delivery, 4 months post delivery

SECONDARY OUTCOMES:
Proportion who progress to the action criteria for effectively managing stress (at baseline not meeting criteria) | Third trimester of pregnancy, 1 month post delivery, and 4 months post delivery
  Assessed by readiness to effectively manage stress each day.
Proportion who progress to the action criteria for eating enough fruits and vegetables (at baseline not meeting criteria) | Third trimester of pregnancy, 1 month post delivery, and 4 months post delivery
  Assessed by readiness to eat at least 5 servings of fruits and vegetables each day.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne D Mauriello, Ph.D., Principal Investigator — Pro-Change Behavior Systems Inc.

REFERENCES:
- [Background] Mauriello L, Dyment S, Prochaska J, Gagliardi A, Weingrad-Smith J. Acceptability and feasibility of a multiple-behavior, computer-tailored intervention for underserved pregnant women. J Midwifery Womens Health. 2011 Jan-Feb;56(1):75-80. doi: 10.1111/j.1542-2011.2010.00007.x. PMID 21323854
- [Background] Prochaska JM, Mauriello L, Dyment S, Gokbayrak S. Designing a health behavior change program for dissemination to underserved pregnant women. Public Health Nurs. 2011 Nov-Dec;28(6):548-55. doi: 10.1111/j.1525-1446.2011.00959.x. Epub 2011 Aug 1. PMID 22092465
- [Derived] Mauriello LM, Van Marter DF, Umanzor CD, Castle PH, de Aguiar EL. Using mHealth to Deliver Behavior Change Interventions Within Prenatal Care at Community Health Centers. Am J Health Promot. 2016 Sep;30(7):554-62. doi: 10.4278/ajhp.140530-QUAN-248. Epub 2016 Jun 16. PMID 26305603